CLINICAL TRIAL: NCT07045922
Title: Effects of Motor-Cognitive Training on Cognitive Performance and Balance in Preschool Children
Brief Title: Motor-Cognitive Training , Cognitive Performance and Balance
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Principal Investigator, Monira Aldhahi, Associate Prof, Princess Nourah Bint Abdulrahman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PNU-5
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-06

CONDITIONS: Coordination Impairment; Children; Balance
MeSH Terms: conditions — Ataxia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor-Cognitive Training Program (Experimental): • Motor-Cognitive Training Program: Game-based physical activities targeting cognitive and motor domains (e.g., running drills, hand skills, stability tasks). Exercises progressed weekly in complexity and duration. Sessions lasted 25-30 minutes, twice weekly.
  Interventions: Behavioral: Motor-Cognitive Training Program; Other: Regular Physical education classes
- Regular Physical education (Other): • Regular PE classes only; no additional physical or motor training permitted.
  Interventions: Other: Regular Physical education classes

INTERVENTIONS:
Behavioral: Motor-Cognitive Training Program — Participants assigned to the intervention group participated in a structured motor-cognitive training program in addition to their regular physical education (PE) classes. The training was designed to integrate physical movement with cognitive engagement in a game-based format, suitable for the preschool age group.
  The program was conducted twice weekly for eight weeks, with each session lasting approximately 25-30 minutes. Activities progressed in complexity over time, incorporating elements of motor planning, executive functioning, and balance control. Sessions consisted of:
  Warm-up phase: Light aerobic activities such as jogging, dynamic stretching, and coordination drills (e.g., knee pulls, toe walking).
  Main training phase: Activities targeting core cognitive-motor domains l
  Arms: Motor-Cognitive Training Program
Other: Regular Physical education classes — Participants in the control group continued with their regularly scheduled physical education (PE) classes as mandated by the school curriculum. They did not receive any additional motor-cognitive or structured exercise training. Furthermore, they were instructed not to engage in any external physical activity programs outside of the regular PE sessions throughout the study duration. This restriction was monitored to ensure group consistency.

SUMMARY:
This RCT design investigates the effects of an 8-week motor-cognitive training program on cognitive performance and balance in preschool-aged children. Participants in the intervention group received structured motor-cognitive activities twice a week in addition to their regular physical education (PE) classes. The control group attended only standard PE classes and was restricted from participating in any other physical activity. Assessments included cognitive testing (Go/No-Go, Tower of Hanoi, and Corsi Block), anthropometric measurements, and static/proprioceptive balance testing. All measurements were conducted pre- and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Typically developing preschool-aged children
* Able to follow basic instructions
* Parental/guardian consent obtained

Exclusion Criteria:

* Diagnosed neurodevelopmental disorders
* Recent musculoskeletal injuries
* Participation in other structured physical activity programs

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive Function Tests | Administered at baseline (pre-intervention) and 8 weeks (post-intervention)
  Evaluates inhibitory control, a core component of executive functioning. Participants are required to respond quickly to target stimuli (e.g., "X") while inhibiting responses to non-target stimuli (e.g., "O"). Measures include:
  Number of correct responses (go trials)
  Number of commission errors (false responses to no-go trials)
  Reaction time (latency) to correct go stimuli
  Duration: ~5 minutes and 40 seconds
Tower of Hanoi Test executive functioning | Baseline and 8 weeks
  Assesses executive functioning, including planning, problem-solving, and cognitive flexibility. Participants solve a visual puzzle by moving disks across pegs, following specific rules. Performance variables include:
  * Number of moves to solution
  * Total task completion time
  * Average time per move
  * Latency to first move (planning time)
Balance Performance | Baseline and 8 weeks
  Balance was assessed using the Sensbalance MiniBoard, a validated interactive platform that captures both static and proprioceptive balance. Two types of balance tasks were used:
  Static Balance Test: Participants were instructed to maintain a stable position on the balance board while keeping a ball centered within a visual target zone on the screen.
  The performance level (%) was calculated using the formula: (1 - Measured Sway Amplitude / Maximum Allowable Sway) × 100, indicating the participant's ability to maintain balance within defined limits.

CONTACTS AND LOCATIONS:
Locations (1):
- Tekirdağ Namik Kemal University, Tekirdağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided